CLINICAL TRIAL: NCT00387608
Title: A Phase 0 Pharmacokinetic, Pharmacodynamic Study of ABT-888, an Inhibitor of Poly (ADP-ribose) Polymerase (PARP), in Refractory Solid Tumors and Lymphoid Malignancies
Brief Title: ABT-888 in Patients With Refractory Solid Tumors or Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 060172; 06-C-0172; NCI-P6890; CDR0000487701; NCT00347633 (obsolete NCT alias)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Leukemia; Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular | interventions — veliparib; Biopsy

INTERVENTIONS:
Drug: veliparib
Other: pharmacological study
Procedure: biopsy

SUMMARY:
RATIONALE: ABT-888 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Collecting and storing samples of blood from patients with cancer to study in the laboratory may help doctors learn more about the ways a patient's body handles the drug.

PURPOSE: This early phase I trial is studying the side effects and best dose of ABT-888 in patients with refractory solid tumors or hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-range at which ABT-888 inhibits poly (ADP-ribose) polymerase (PARP) in tumor samples and in peripheral blood mononuclear cells (PBMCs) in patients with refractory solid tumors or lymphoid malignancies.
* Determine the pharmacokinetics of ABT-888.
* Determine the time course of PARP inhibition in PBMCs by ABT-888.

Secondary

* Determine the safety of administering 1 dose of ABT-888 in these patients.

OUTLINE: This is a dose-finding study.

Patients receive oral ABT-888 once on day 1.

Cohorts of 3 patients receive escalating doses of ABT-888 until significant tumor poly (ADP-ribose) polymerase (PARP) inhibition is observed in 3 of 3 patients at 2 dose levels. Significant PARP inhibition is defined as ≥ 0.69 reduction on the log scale in poly (ADP-ribose) level from baseline to 3-6 hours after ABT-888 administration (with 90% confidence that it is not due to chance variation).

Patients undergo peripheral blood collection at baseline and periodically after ABT-888 administration for PARP inhibition, pharmacokinetic, and pharmacodynamic studies. Once significant PARP inhibition is observed in 1 of 3 patients, subsequently enrolled patients also undergo tumor biopsy* at baseline and 3-6 hours or 21-27 hours after ABT-888 administration to determine PARP inhibition in tumor tissue.

NOTE: *Patients with chronic lymphocytic leukemia undergo peripheral blood collection instead of biopsy.

After completion of ABT-888 administration, patients are followed for 7 days.

PROJECTED ACCRUAL: A total of 23 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignancy, meeting 1 of the following criteria:

  * Solid tumor that is refractory to ≥ 1 line of standard treatment OR for which no standard therapy is available

    * Must have ≥ 1 lesion amenable to percutaneous biopsy (for solid tumor patients enrolled after the initial phase of the study)
  * Chronic lymphocytic leukemia (CLL) or follicular lymphoma with no current indication for standard therapy OR disease that has failed ≥ 1 line of standard therapy
* No disease-associated symptoms requiring immediate therapy or other interventions
* Must be willing to undergo tumor biopsies* after the initial phase of the study NOTE: *Patients with CLL undergo peripheral blood collection instead of biopsy
* No primary brain tumors, brain metastases, or leptomeningeal disease

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 or Karnofsky PS 60-100%
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine < 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* INR ≤ 1.4
* PTT ≤ 36 seconds
* Calcium (corrected) normal
* Magnesium < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 30 days after study completion
* No history of seizures
* No evidence of bleeding diathesis
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmias
* No psychiatric illness or social situations that would limit study compliance

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior radiation therapy or surgery and recovered
* At least 2 weeks since other prior therapy and recovered
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent lung, liver, or mediastinal lymph node biopsies
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change in tumor poly (ADP-ribose) (PAR) levels from baseline to 3-6 hours after ABT-888 administration
Pharmacokinetics

SECONDARY OUTCOMES:
Safety of administering 1 dose of ABT-888
Changes in PAR levels in peripheral blood mononuclear cells from baseline to after ABT-888 administration

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, MD, Principal Investigator — NCI - Medical Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States

REFERENCES:
- [Result] Kummar S, Kinders R, Gutierrez ME, Rubinstein L, Parchment RE, Phillips LR, Ji J, Monks A, Low JA, Chen A, Murgo AJ, Collins J, Steinberg SM, Eliopoulos H, Giranda VL, Gordon G, Helman L, Wiltrout R, Tomaszewski JE, Doroshow JH. Phase 0 clinical trial of the poly (ADP-ribose) polymerase inhibitor ABT-888 in patients with advanced malignancies. J Clin Oncol. 2009 Jun 1;27(16):2705-11. doi: 10.1200/JCO.2008.19.7681. Epub 2009 Apr 13. PMID 19364967